CLINICAL TRIAL: NCT06526494
Title: Metformin and Vascular Function in Prediabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: Diana Jalal (Other)
Responsible Party: Sponsor-Investigator, Diana Jalal, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202403617
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: PreDiabetes
Keywords: vascular function; metformin; prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Participants will receive metformin 850 mg PO once a day for 2 weeks. After 2 weeks, participants will receive metformin 1700 mg PO once a day for the remaining 10 weeks.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Patients will receive placebo pill identical in appearance and taste to the supplement
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — Oral ingestion for 12 weeks
  Arms: Metformin
Other: Placebo — Oral placebo for 12 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate whether metformin improves vascular function in individuals with prediabetes. The main questions it aims to answer are:

1. Does metformin improve large conduit artery endothelial function in individuals with prediabetes?
2. Does metformin improve microvascular endothelial function in individuals with prediabetes?

Researchers will compare metformin to a placebo to see if metformin improves vascular function in prediabetes.

The trial duration is 12 weeks. Participants will take metformin or a placebo once a day for 2 weeks. After 2 weeks, participants will take metformin or a placebo twice a day for the remaining 10 weeks. There will be a screening visit, two baseline visits, a 4-week safety visit, and two 12-week end-of-study visits. Adherence will be calculated from pill count and adverse events will be quantified via a questionnaire.

DETAILED DESCRIPTION:
Prediabetes affects approximately 98 million people in the United States and significantly elevates the risk of cardiovascular disease (CVD) and progression to type-2 diabetes. Endothelial dysfunction, characterized by reduced nitric oxide bioavailability, is a key subclinical risk factor contributing to the increased CVD risk in prediabetes. Additionally, endothelial dysfunction exacerbates insulin resistance and hyperglycemia, further elevating the likelihood of progression to overt diabetes. Thus, targeting endothelial dysfunction in prediabetes presents a strategic opportunity to mitigate the risks of both CVD and overt diabetes.

Hyperglycemia-induced reactive oxygen species (ROS) generation reduces nitric oxide bioavailability, driving endothelial dysfunction in prediabetes. Therefore, interventions that lower hyperglycemia could decrease ROS production, enhance nitric oxide bioavailability, and improve endothelial function in prediabetes. Metformin, a first-line anti-diabetic agent, lowers hyperglycemia by reducing hepatic glucose output and enhancing insulin-mediated glucose uptake. Despite its established vascular benefits in diabetes, the effects of metformin on endothelial function in prediabetes remain unexplored.

This study will enroll 30 individuals in a randomized, double-blind, placebo-controlled clinical trial utilizing innovative methodologies to elucidate the vascular benefits of metformin in prediabetes. Specifically, the investigators will assess 1) large conduit artery endothelial function, and 2) cutaneous microvascular endothelial function in prediabetes. By investigating these mechanisms, the investigators aim to provide critical insights into metformin's potential to reduce CVD risk and prevent the progression to diabetes in individuals with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Prediabetes defined as an HbA1c between 5.7% and 6.4%
* Able to provide informed consent

Exclusion Criteria:

* Current use of metformin or metformin use within the past 12 months
* Current use of medicated contraindicated for use with metformin
* Current use of vitamin C supplement
* Current smoker or quit smoking within the last 6 months
* Pregnant, breastfeeding, planning to become pregnant, or unwilling to use adequate birth control
* Uncontrolled hypertension (Systolic blood pressure >140 mmHg)
* Body Mass Index > 40 kg/m2
* History of diabetes, myocardial infarction, heart failure, liver disease, or chronic kidney disease (estimated glomerular filtration rate < 45 ml/min/1.73m2)
* History of lactic acidosis
* History of alcohol abuse
* Severe infection within the last 30 days
* Immunosuppressive therapy within the past year
* Life expectancy < 1 year
* Allergy to metformin, nitroglycerin, sodium nitroprusside, ringer's lactate
* Study compliance: Unwilling to fast overnight, have an intravenous catheter placed, take a study drug for 12 weeks, or visit Iowa campus 6 times within a 12-16 week period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Macrovascular endothelial function | 12 weeks
  Brachial artery flow-mediated dilation

SECONDARY OUTCOMES:
Microvascular endothelial function | 12 weeks
  Cutaneous microvascular dilation

CONTACTS AND LOCATIONS:
Overall Officials: Diana I Jalal, MD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: No